CLINICAL TRIAL: NCT01460719
Title: A Phase I, Open-Label, Multicenter Clinical Trial to Evaluate the Safety and Immunogenicity of V212/Inactivated Varicella-Zoster Virus (VZV) Vaccine in Adults With Hematologic Malignancies Receiving Treatment With Anti-CD20 Monoclonal Antibodies
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Inactivated Varicella-Zoster Virus (VZV) Vaccine in Adults With Hematologic Malignancies (HM) Receiving Treatment With Anti-Cluster of Differentiation (CD) 20 Monoclonal Antibodies (V212-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V212-013; V212-013 (Other: Merck Protocol Number); 2011-003153-25 (EudraCT Number)
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- V212 (Experimental): Participants receive V212 as a 0.5 mL subcutaneous injection in a four-dose regimen, approximately 30 days apart, preferably in the deltoid area of the arm, alternating arms for each dose.
  Interventions: Biological: V212

INTERVENTIONS:
Biological: V212 — V212 viral antigen for HZ
  Other Names: Inactivated Varicella-Zoster (VZV) vaccine

SUMMARY:
An open-label, multicenter study to evaluate the safety and immunogenicity of inactivated VZV vaccine (V212) in participants with hematologic malignancies (HM) who are currently receiving anti-CD20 monoclonal antibodies. The primary hypothesis is that vaccination with V212 vaccine will elicit significant VZV-specific immune responses at ~28 days after vaccination 4. The statistical criterion for significance requires that the lower bound of the 2-sided 90% confidence interval of the geometric mean fold rise in immune response in V212 recipients is >1.0.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a HM and is receiving treatment with anti-CD20 monoclonal antibodies and is not likely to undergo hematopoietic cell transplant (HCT).
* Has a predicted life expectancy of ≥ 12 months.
* Has prior history of varicella or antibodies to VZV due to exposure to the disease in a country where the disease is common.
* All female participants of childbearing potential must have a negative serum or urine pregnancy test.

Exclusion Criteria:

* A history of allergic reaction to any vaccine component (including gelatin) or an anaphylactic/anaphylactoid reaction to neomycin.
* Prior history of HZ within 1 year of enrollment.
* Prior receipt of any varicella or zoster vaccine.
* Participant is pregnant or breastfeeding or expecting to conceive within the period of 2 weeks prior to enrollment throughout 6 months after last vaccination dose.
* Any live virus vaccine administered or scheduled in the period from 4 weeks prior to Dose 1 through 28 days postvaccination dose 4.
* Any inactivated vaccine administered or scheduled within the period from 7 days prior to, through 7 days following, any dose of study vaccine.
* Participant is currently participating or has participated in a study with an investigational anti-CD20 monoclonal antibody within 3 months of signing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2012-09-25 (Actual); Study Completion 2012-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Parrino J, McNeil SA, Lawrence SJ, Kimby E, Pagnoni MF, Stek JE, Zhao Y, Chan IS, Kaplan SS. Safety and immunogenicity of inactivated varicella-zoster virus vaccine in adults with hematologic malignancies receiving treatment with anti-CD20 monoclonal antibodies. Vaccine. 2017 Mar 27;35(14):1764-1769. doi: 10.1016/j.vaccine.2016.10.055. Epub 2017 Mar 3. PMID 28268074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 88 participants were screened and 80 were enrolled.
Groups:
- V212: Participants received V212 as a 0.5 mL subcutaneous injection in a four-dose regimen, approximately 30 days apart, preferably in the deltoid area of the arm, alternating arms for each dose
Period: Overall Study
Arm/Group | V212
Started | 80
Vaccination 1 (Day 1) | 80
Vaccination 2 (~Day 30) | 78
Vaccination 3 (~Day 60) | 78
Vaccination 4 (~Day 90) | 78
Completed | 78
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | V212
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) of the VZV-specific Immune Responses Measured by VZV Interferon-gamma (IFN-γ) Enzyme-linked Immunospot (ELISPOT)
Description: The VZV ELISPOT assay detects IFN-γ-secreting, VZV-specific cells from peripheral blood mononuclear cells (PBMCs). The unit of measure of the assay is ELISPOT cell count / 10^6 PBMCs, and is expressed as geometric mean count (GMC). The GMFR is GMC at ~28 days after Vaccination 4 / GMC on Day 1.
Time Frame: Prevaccination (Day 1) and ~28 days after Vaccination 4 (~Day 118)
Population: Vaccinated participants having valid results at Baseline (Day 1) and/or at ~28 days after Vaccination 4.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | V212
Number analyzed (Participants) | 78
Ratio | 4.34 [3.01 to 6.24]
Statistical Analysis 1: Comparison: V212; Test type: Other — The statistical criterion for significance requires that the lower bound of the 2-sided 90% confidence interval of the GMFR is >1.0; p < 0.001, Single longitudinal regression model; Adjustments made for pre-vaccination values

2. Primary Outcome: Percentage of Participants With an Adverse Event
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the product is also an adverse experience. The percentage of participants with any AE was summarized.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All enrolled participants
Measure: Number; unit: Percentage of participants
Arm/Group | V212
Number analyzed (Participants) | 80
Percentage of participants | 85.0

3. Primary Outcome: Percentage of Participants With an Injection-site Adverse Event
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the product is also an adverse experience. The percentage of participants with any injection-site AE was summarized.
Time Frame: Up to 5 days after any vaccination
Population: All enrolled participants
Measure: Number; unit: Percentage of participants
Arm/Group | V212
Number analyzed (Participants) | 80
Percentage of participants | 43.8

4. Primary Outcome: Percentage of Participants With a Systemic Adverse Event
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the product is also an adverse experience. The percentage of participants with any systemic AE was summarized.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All enrolled participants
Measure: Number; unit: Percentage of participants
Arm/Group | V212
Number analyzed (Participants) | 80
Percentage of participants | 73.8

5. Primary Outcome: Percentage of Participants With a Serious Adverse Event
Description: A serious AE (SAE) is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs an inpatient hospitalization, is a congenital anomaly or birth defect, is an overdose, is a cancer, or is another important medical event. The percentage of participants with any SAE was summarized.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All enrolled participants
Measure: Number; unit: Percentage of participants
Arm/Group | V212
Number analyzed (Participants) | 80
Percentage of participants | 15.0

6. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A serious AE (SAE) is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs an inpatient hospitalization, is a congenital anomaly or birth defect, is an overdose, is a cancer, or is another important medical event. The percentage of participants with any SAE that was deemed by the investigator to be possibly, probably, or definitely related to study vaccine was summarized.
Time Frame: Up to ~28 days after Vaccination 4 (~Day 118)
Population: All enrolled participants
Measure: Number; unit: Percentage of participants
Arm/Group | V212
Number analyzed (Participants) | 80
Percentage of participants | 1.3

7. Primary Outcome: Percentage of Participants With Study Vaccination Withdrawn Due to an Adverse Event
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the product is also an adverse experience. The percentage of participants with study vaccine withdrawn due to an AE was summarized.
Time Frame: Up to Vaccination 4 (~Day 90)
Population: All enrolled participants
Measure: Number; unit: Percentage of participants
Arm/Group | V212
Number analyzed (Participants) | 80
Percentage of participants | 1.3

ADVERSE EVENTS:
Time Frame: Up to Day 140
Description: All participants who received at least one dose of V212
Arm/Group | V212
All-Cause Mortality (participants affected / at risk) | 1/80
Serious Adverse Events (participants affected / at risk) | 12/80
Other Adverse Events (participants affected / at risk) | 67/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212 (N=80)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Salmonellosis (Infections and infestations) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal squamous cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212 (N=80)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (7)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (13)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Feeling hot (General disorders) | 1 (2)
Injection site erythema (General disorders) | 25 (54)
Injection site haematoma (General disorders) | 2 (2)
Injection site movement impairment (General disorders) | 1 (2)
Injection site pain (General disorders) | 26 (57)
Injection site paraesthesia (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 5 (9)
Injection site rash (General disorders) | 2 (2)
Injection site swelling (General disorders) | 21 (49)
Malaise (General disorders) | 1 (1)
Mucosal dryness (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 20 (27)
Spinal pain (General disorders) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Acariasis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Trichophytosis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral tracheitis (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 6 (10)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (9)
Hypoaesthesia (Nervous system disorders) | 2 (3)
Migraine (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (2)
Rash vesicular (Skin and subcutaneous tissue disorders) | 5 (5)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (2)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.